CLINICAL TRIAL: NCT03858881
Title: Building Evidence-Based Supports for Teens Via Technology
Acronym: BEST-TECH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Limbix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1337335-2
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be partly blind to condition =. A computer-based survey will randomize participants into one of three conditions: an online mindset program, an online control program, or a virtual reality program. If a participant is randomized into one of the first 2 programs, the participant will know that s/he is not assigned to the VR program, but neither the experimenter nor the participant will be aware of which of the two computer-based programs s/he is completing. However, both participants and the experimenter leading the study visit will be aware of whether he participant was allocated to the VR condition (specific equipment set-up is required). The experimenters leading the study visits will be trained RAs not involved in data analysis. The study PI will remain blind to participants' condition assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PROJECT PERSONALITY (Active Comparator)
  Interventions: Behavioral: PROJECT PERSONALITY
- VR PERSONALITY PROJECT (Experimental)
  Interventions: Behavioral: VR PERSONALITY PROJECT
- SHARING FEELINGS PROGRAM (Placebo Comparator)
  Interventions: Behavioral: SHARING FEELINGS PROGRAM

INTERVENTIONS:
Behavioral: PROJECT PERSONALITY — PROJECT PERSONALITY is self-administered by youth via Qualtrics and is 30 minutes in duration. The intervention includes five elements: 1. An introduction to the brain, including a lesson on neuroplasticity (how and why our behaviors are controlled by thoughts and feelings in the brains, which have potential for change); 2. Testimonials from older youths who describe their views that people's traits are malleable, given the brain's plasticity; 3. Additional vignettes written by older youths, describing times when they used "growth mindsets" to persevere through social and emotional setbacks; 4. A summary of selected scientific studies suggesting that personality can, and often does, change in positive ways over time; and 5. An exercise in which the participants write notes to younger students, drawing on scientific information to describe the malleability of people's personal traits
  Other Names: Web-based growth mindset intervention
  Arms: PROJECT PERSONALITY
Behavioral: VR PERSONALITY PROJECT — The VR PERSONALITY PROJECT contains similar elements as PROJECT PERSONALITY, including a lesson on neuroplasticity; testimonials from older youths; information about research on the malleability of personal traits; and an exercise wherein the participant provides advice to a student in the VR environment who has experienced a peer-related setback. Content is delivered by characters in the VR environment (hired/filmed actors) who guide youths through the program, providing scientific information and personal stories. Completion time is 30-40 minutes. The key difference between the VR and web-based mindset intervention is the delivery system, and by extension the level of immersion each program offers. The VR program is designed to be immersive, fun and interactive; youth choose to speak to various scientists and students within the VR environment and navigate themselves from scene to scene. In the online program, participants automatically view a series of text-based activities.
  Other Names: Virtual reality growth mindset intervention
  Arms: VR PERSONALITY PROJECT
Behavioral: SHARING FEELINGS PROGRAM — The web-based supportive therapy (ST) intervention, called the Sharing Feelings Program, is delivered via Qualtrics, self-administered by youth, and 30 minutes in duration. It aims to encourage youths to identify and express feelings to close others and does not teach specific skills or beliefs. It is designed to control for nonspecific aspects of intervention, including engagement in a technology-based program. It mirrors the web-based growth mindset intervention as closely as possible, including vignettes written by older youths who describe times when they benefited from sharing their feelings with friends or family.
  Other Names: Web-based supportive therapy intervention
  Arms: SHARING FEELINGS PROGRAM

SUMMARY:
Major depression (MD) is the leading cause of disability in youth, with a global economic burden of >$210 billion annually. However, up to 70% of youth with MD do not receive services. Even among those who do access treatment, 30-65% fail to respond, demonstrating a significant need for more potent, accessible interventions for adolescent depressive symptoms and disorders.

The goal of this project is to assess the acceptability and effectiveness of a novel, single-session, virtual reality-based depression intervention-the VR Personality Project-teaching growth mindset: the belief that personal behaviors and characteristics, such as depressive symptoms, are malleable rather than fixed. In a previous trial, a single-session growth mindset intervention significantly reduced depressive symptoms in high symptom-adolescents; however, this intervention did not benefit all adolescents uniformly. For instance, the intervention reduced depression in adolescents who reported post-intervention increases in perceived control, but it did not lead to significant depression reductions in adolescents who reported small or no increases in perceived control. Thus, the VR Personality Project was designed to systematically target and increase adolescents' perceived control by offering a more immersive, active, and user-directed intervention experience than the web-based SSI can provide. By targeting an identified predictor of intervention response, the VR Personality Project may be lead to larger reductions in depression than the existing web-based mindset SSI.

To test this possibility, adolescents with elevated depressive symptoms or at high risk for depressive symptoms (N=159; ages 12-16) will be randomized to one of three intervention conditions: the VR Personality Project; the web-based growth mindset SSI tested previously; or an active control SSI, also tested previously. Adolescents and their parents will report on their depression symptoms, perceived control, and related domains of functioning at pre-intervention, post-intervention, and at three- and nine-month follow-ups. We predict that the VR and web-based SSIs will both lead to larger reductions in adolescent symptoms relative to the control SSI. Additionally, we predict that the VR-based SSI will lead to larger reductions in depression than the online SSI, and that these symptom reductions will be mediated by increases in adolescents' perceived control. Results may identify a particularly potent, mechanism-targeted, brief intervention for adolescent depression.

DETAILED DESCRIPTION:
Psychiatric disorders are the leading cause of disability worldwide, and 40.5% of this burden is attributable to major depression (MD). Rates of MD increase markedly in adolescence, with nearly 20% of youth experiencing MD between ages 12 and 18. Adolescent-onset MD accounts for 66% of lifetime MD cases and predicts interpersonal problems, substance abuse, and a 20-fold increased risk for attempting suicide. Despite this early onset and protracted course, up to 70% of US adolescents with MD do not receive services. Even among those who do access treatment, 30-65% fail to respond. These findings highlight the urgent need for more potent and accessible MD interventions for adolescents.

Emerging work suggests that single-session interventions (SSIs) may increase accessibility of youth MD interventions. SSIs include core elements of comprehensive, evidence based treatments, but their brevity makes them easier to disseminate to diverse settings. Indeed, SSIs can successfully treat youth psychiatric problems: In a meta-analysis of 50 RCTs, it has been found that SSIs reduced youth mental health difficulties of multiple types (mean g=0.32), including self-administered SSIs (e.g., web-based SSIs; mean g=0.32). One SSI, in particular, has been shown to reduce adolescent MD symptoms: the growth mindset (GM) SSI, a web-based program teaching the belief that personal traits are malleable, which has prevented and reduced adolescent MD in recent RCTs. For example, in a recent RCT conducted by the principal investigator on the proposed study, the GM SSI led to post-intervention increases in adolescents' perceived control over behavior (d=.34, p<.001) and emotions (d=.19, p=.03) relative to a comparison (supportive therapy, or ST) SSI. The GM SSI also predicted steeper 9-month declines in youth depression symptoms per parent (B=-.99, p=.047) and adolescent reports (B=-1.37, p=.03), based on mixed-effects linear models.

However, it is notable that the GM SSI does not reduce depression in all adolescents. For instance, the intervention reduced depression in adolescents who reported post-intervention increases in perceived control over behaviors and emotions, but it did not lead to significant depression reductions in adolescents who reported small or no increases in perceived control. Thus, the potency of GM SSIs for adolescent depression has yet to be optimized. Such potency may be advanced by developing new iterations of the growth mindset intervention, which are designed to more systematically target predictors and mediators of clinical outcomes, such as perceived control. Such efforts may increase the promise of growth mindset interventions to produce greater symptom reductions for a larger proportion of youth experiencing distress.

Accordingly, the goal of the present study is to test the acceptability and effectiveness of a novel, single-session virtual reality-based growth mindset intervention-the VR Personality Project-for depressive symptoms in adolescents. The VR Personality Project was designed to systematically target and increase adolescents' sense of agency and perceived control by offering a more immersive, active, and user-directed intervention experience than the previously-tested web-based SSI can provide. By targeting an identified predictor and mechanism of intervention response, the VR Personality Project may produce larger reductions in depression than the existing web-based mindset SSI. Thus, this intervention may represent a mechanism-targeted, efficient strategy for reducing for adolescent depression--one that is both relatively affordable (less than $100 for any commercially-available VR headset, a fraction of the cost of long-term psychotherapy) and engaging to adolescents experiencing mood-related distress.

There are four specific study aims for this research:

AIM 1: Replication of past research. Our first aim is to replicate past research suggesting that single-session growth mindset interventions can significantly reduce depressive symptoms in at-risk adolescents. We hypothesize that adolescents who participate in a growth mindset intervention (web-based OR virtual reality-based) will show larger reductions in depression symptoms from baseline (pre-intervention) through the 9-month follow-up assessment, compared to adolescents who receive an active, web-based control program.

AIM 2: Evaluation of new virtual reality intervention, including a comparative efficacy study. Our second aim is to evaluate whether the new virtual reality-based growth mindset intervention (the VR Personality Project) can reduce depressive symptoms in adolescents, both relative to an active control program and relative to the previously tested web-based growth mindset intervention. We hypothesize that adolescents who participate in the virtual reality-based growth mindset intervention will show larger reductions in depressive symptoms from baseline (pre-intervention) through the 9-month follow-up assessment, compared to adolescents who receive the web-based growth mindset intervention AND adolescents who receive the active web-based control program.

AIM 3: Testing mediation through perceived control. The VR Personality Project was explicitly designed to target and increase adolescents' perceived control by offering a more immersive, active, and user-directed intervention experience than the the web-based growth mindset SSI can provide. Thus, the third goal of this study is to examine whether the VR Personality Project does, in fact, reduce adolescent depressive symptoms by eliciting proximal increases in perceived control. We hypothesize that the VR Personality Project will lead to larger increases in perceived control than either web-based intervention from pre- to post-intervention, and that these increases will mediate subsequent reductions in adolescent depression across the follow-up period.

AIM 4: Gauge the relative acceptability and feasibility of the VR intervention. Adolescents' perceptions of any intervention can impact completion rates, program engagement, and ultimately intervention effectiveness. Thus, an additional aim of this research is to examine whether adolescents view the VR Personality Project as more engaging, helpful, and interesting than the web-based growth mindset intervention or the web-based control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Youth is between the ages of 12-16 years (inclusive) at the time of study enrollment
* Youth has one parent or legal guardian willing to participate in the study (i.e., to be present for the lab visit and to complete questionnaires throughout the study period)
* Youth speaks English well enough to complete online or virtual reality-based intervention activities, which are available in English only
* Indication of elevated risk for youth depression. This criterion may be met in one of two ways (or both ways): (a) The adolescent exhibits elevations in depressive symptoms (subclinical or greater symptom elevations, corresponding to 80th percentile or higher, based on parent-report CDI 2 conducted an initial phone screen); (b) The adolescent received treatment for depression within the previous 2 years (depression tends to recur, so past treatment receipt indicates elevated risk). Past treatment receipt will be assessed via parent report at the time of the phone screen.

Exclusion Criteria:

* Intellectual disability, as this may undermine comprehension of intervention materials
* Adolescent is non-English speaking, as the virtual reality and online interventions are available in English only;
* Adolescent was hospitalized or received residential/inpatient treatment for suicide attempt or self-harming behaviors within the past 2 months, as the interventions being tested in this study are not designed for adolescents with acute medical and/or psychiatric treatment needs

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Depression Inventory - 2 (Youth Report) | Baseline to 3- and 9-month follow-up
  Change in youth reported depressive symptoms, total score derived from 28-item CDI-2. Scores range from 0-56, with higher scores indicating higher levels of depression.
Change in Children's Depression Inventory - 2 (Parent Report) | Baseline to 3- and 9-month follow-up
  Parent reported youth depressive symptoms, total score derived from 17-item parent-report version of CDI-2. Scores range from 0-54, and higher scores indicate greater youth depression severity.

SECONDARY OUTCOMES:
Change in Screen for Anxiety Related Disorders (Youth Report) | Baseline to 3- and 9-month follow-up
  Youth reported anxiety symptoms, total score derived from 41-item SCARED. Scores range from 0 to 82. Higher scores indicate greater anxiety severity.
Change in Screen for Anxiety Related Disorders (Parent Report) | Baseline to 3- and 9-month follow-up
  Change in parent reported youth anxiety symptoms, total score derived from 41-item SCARED-P. Scores range from 0 to 82. Higher scores indicate greater anxiety severity.
Change in Perceived Control Scale for Children | Baseline to immediate post-intervention, 3-month, and 9-month follow-ups.
  Youth-reported perceptions of control over behavioral responses to setbacks. Total score is derived from the sum of all items in the 24-item scale (range: 0 - 72), with higher scores reflecting higher levels of perceived control.
Change in Secondary Control Scale for Children | Baseline to immediate post-intervention, 3-month, and 9-month follow-ups.
  Youth-reported perceptions of control over emotional responses to setbacks. Total score is derived from the sum of all items in the 20-item scale (range: 0 - 60), with higher scores reflecting higher levels of perceived control.
Change in UCLA Loneliness Scale | Baseline to immediate post-intervention, 3-month, and 9-month follow-ups.
  The ULS is a widely used self-report scale of loneliness in adolescents. The 20-item version will be used here. Adolescents rate how often they experience loneliness in various contexts (e.g., 'how often do you feel part of a group of friends?' 'How often do you feel there is no one you can turn to?'). Higher scores indicate higher levels of loneliness. Scores range from 0-60.
Change in Attitudes Toward Therapy Scale - Youth | Baseline to immediate post-intervention, 3-month, and 9-month follow-ups.
  One-item measure used to assess youths' perceptions that therapy/counseling would be useful in reducing emotional or behavioral difficulties, rated on a 0-10 scale (total score range: 0-10). Higher scores indicate stronger beliefs that therapy may help reduce mental health problems, whereas lower scores indicate weaker beliefs that therapy may help reduce mental health problems.
Change in Attitudes Toward Therapy Scale - Parent | Baseline to 3-month and 9-month follow-ups.
  One-item measure used to assess parents' perceptions that therapy/counseling would be useful in reducing their child's emotional or behavioral difficulties, rated on a 0-10 scale (total score range: 0-10). Higher scores indicate stronger beliefs that therapy may help reduce mental health problems, whereas lower scores indicate weaker beliefs that therapy may help reduce mental health problems.
Change in Beck Hopelessness Scale-4 | Baseline to immediate post-intervention, 3-month, and 9-month follow-ups.
  Respondents (youths) report agreement with 4 items indicating levels of hopelessness about the future. Higher summed scores reflect greater levels of hopelessness, and scores range from 0-12.
Change in Implicit Theories of Personality Questionnaire, youth-report | Baseline to immediate post-intervention, 3-month, and 9-month follow-ups
  Respondents rate the extent of their agreement with three statements linked to the malleability of personality, using a 1-to-7 Likert scale (e.g. "Your personality is something about you that you can't change very much"). Higher mean scores on these three items indicate a stronger fixed personality mindset, a lower scores, a stronger growth personality mindset (range: 1-7).

OTHER OUTCOMES:
Change in Implicit Theories of Personality Questionnaire, parent-report | Baseline to 3-month and 9-month follow-ups
  Respondents rate the extent of their agreement with three statements linked to the malleability of personality, using a 1-to-7 Likert scale (e.g. "Your personality is something about you that you can't change very much"). Higher mean scores on these three items indicate a stronger fixed personality mindset, a lower scores, a stronger growth personality mindset (range: 1-7).
Change in Brief Symptom Inventory-18 | Baseline to 3-month and 9-month follow-ups
  The Brief Symptom Inventory-18 (BSI-18) assesses self reported parent psychopathology and distress. Adult respondents rate endorsement of 18 physical and emotional complaints on a 0-4 Likert scale. The total sum score yields an additional total distress score (range: 0-72). Higher scores indicate higher levels of overall psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

REFERENCES:
- [Derived] Schleider JL, Mullarkey MC, Weisz JR. Virtual Reality and Web-Based Growth Mindset Interventions for Adolescent Depression: Protocol for a Three-Arm Randomized Trial. JMIR Res Protoc. 2019 Jul 9;8(7):e13368. doi: 10.2196/13368. PMID 31290406